CLINICAL TRIAL: NCT02568800
Title: Prolonged Infusion Cefepime and Nosocomial Infections
Acronym: PICNIC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-0392
Record Dates: First submitted 2015-10-02; First posted 2015-10-06 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Urinary Tract Infection; Respiratory Tract Infection
MeSH Terms: conditions — Urinary Tract Infections; Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolonged Cefepime Infusion (Experimental): Cefepime infusions should last 4 hours at least
  Interventions: Drug: Prolonged Cefepime Infusion
- Usual Cefepime Infusion (Active Comparator): Cefepime infusion should last no more than 30 minutes
  Interventions: Drug: Usual Cefepime Infusion

INTERVENTIONS:
Drug: Prolonged Cefepime Infusion — Cefepime infusion should last at least 4 hours with the aide of an infusion bomb
  Other Names: Estended Cefepime Infusion
  Arms: Prolonged Cefepime Infusion
Drug: Usual Cefepime Infusion — Cefepime infusion occurs directly without the aide of an infusion bomb, lasting roughly thirty minutes
  Other Names: Regular Cefepime Infusion
  Arms: Usual Cefepime Infusion

SUMMARY:
It is advocated that prolonged infusion of beta-lactamic antibiotics provides better bactericidal effect. The aim of the present study is to randomize patients a to extended cefepime infusion regimen (lasting four hours) or to a usual infusion regimen (not lasting more than thirty minutes) and evaluate the clinical efficacy of this theoretical pharmacokinetic advantage.

DETAILED DESCRIPTION:
Introduction: it has been proved that the main determinant for microbiological cure gram-negative infections treated with cefepime is the time above minimal inhibitory concentration (T>MIC). Although this particular pharmacokinetic property have never been proved in clinical trials utilizing cefepime, intervention studies with other betalactamic antibiotics, such as pipercillin-tazobactam, showed clinical benefit.

Objective: to evaluate if prolonged infusion (lasting 4 hours) with cefepime translate into better clinical outcomes.

Methods: the investigators aim to conduct an open-label, unique-centered, randomized controlled trial using cefepime in prolonged infusions in patients being treated for urinary or respiratory tract infections. Patients developing these infections after 72 hours of hospital admission, requiring the use of broader spectrum antibiotics after clinical failure or isolating gram-negative bacteria from adequate sample sensible to cefepime will be enrolled. The use of a second antibiotic such as clindamycin, vancomycin or metronidazole will be allowed.

Interventions: the investigators aim to randomize 134 patients to two different treatment arms, the intervention arm who will receive the medication in a four hour lasting infusion, and the active control arm who will receive the medication in a 30 minutes lasting infusion. The randomization will be conducted in blocks of ten patients each, and it will be balance according to the patients age (older or younger than 65 years old) and presence of SIRS criteria.

ELIGIBILITY:
Inclusion Criteria:

* Urinary tract infection after 48-72 hours of hospital stay
* Respiratory tract infection after 48-72 hours of hospital stay
* Catheter related urinary tract infection after 48-72 hours of hospital stay
* Urinary or respiratory infections not responding to a narrower spectrum antibiotic
* Isolation of bacteria sensible to cefepime in blood, urine or sputum in a clinical context of infection

Exclusion Criteria:

* Glomerular filtration rate lower than 30 ml.min/1,73m²
* ICU admission for at least 72 hours before randomization
* Neutrophil count lower than 1000 cels per mm³
* Hematologic malignancy, bronchiectasis and cystic fibrosis
* Patients allergic to cefepime
* Concomitant treatment to another infectious disease
* Central nervous system, cutaneous or intrabdominal infections
* Solid organ transplantation
* HIV with a cluster differentiation 4 (CD4) lower than 100 cels per mm³

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-03 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Death | 30 days
  Death in 30 days since randomization

SECONDARY OUTCOMES:
Death | 14 days
  Death in 14 days since randomization
Duration of hospital stay | 30 days since randomization
  Duration of hospital stay
Intensive care unit (ICU) admission | 30 days since randomization
  Intensive care necessity for any reason
Duration of intensive care unit (ICU) stay | 30 days since randomization
  Number of days when intensive care was considered necessary
Treatment change | 3 days after randomization
  Treatment change required based com clinical or microbiological data
Treatment success | 30 days since randomization
  Patient reaching the completion until it end with infection resolution
Time to clinical stability | 3 days
  Time required for patient to reach the normalization of all following vital signs: that is, body temperature lower than 37,9 degrees celsius, a cardiac rate lower than 100 beats per minute and a respiratory rate lower than 25 respiratory movements per minute and peripheral oxygen saturation higher than 91% with low oxygen requirement (that is 4 liters per minute delivered by nasal canula)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Sprinz, Principal Investigator — Hospita de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil